CLINICAL TRIAL: NCT04716660
Title: Changes in Sensory Block Level During a Programmed Intermittent Epidural Bolus Regimen for Labor Analgesia: an Observational Cohort Study
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21-01
Record Dates: First submitted 2021-01-12; First posted 2021-01-20 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Labor Pain
Keywords: programmed intermittent epidural bolus; epidural analgesia; labor epidural; sensory block
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women receiving epidural analgesia for labor
  Interventions: Other: Sensory block level check

INTERVENTIONS:
Other: Sensory block level check — Patients will have their sensory block level checked multiple times following administration of their epidural bolus for labor analgesia.

SUMMARY:
Epidural analgesia is widely used for managing pain during labor. The programmed intermittent epidural bolus (PIEB) technique has been shown to produce less consumption of local anesthetics, better sensory block, less motor block, and increased maternal satisfaction than other epidural analgesia techniques. Despite all benefits from PIEB, such practice has been associated with high sensory block levels. Therefore, assessment of the sensory block level is an essential component of clinical safety. The lack of a standardized technique and timing to assess the sensory block level can lead to inappropriate management. The purpose of this study is to investigate the changes in block level over time, during cycles of a PIEB regimen. The investigators hypothesize that these levels will be highest soon after the PIEB bolus and lowest preceding the subsequent PIEB bolus. The investigators also want to investigate a possible correlation between these changes in sensory block levels and motor block, pain scores, and rescue bolus of local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* women admitted to the Labor and Delivery unit at Mount Sinai Hospital that request and have no contraindications to receive epidural analgesia
* 18 years old or more
* capable of understanding and signing the written informed consent
* have no language barrier to respond to the level of sensory block assessment
* and have no conditions that could compromise the body sensitivity to cold.

Exclusion Criteria:

* unintentional dural puncture during labour epidural placement
* do not achieve adequate pain control 20 minutes after the loading dose (numeric rating scale (NRS)>1 on a 0-10 NRS),
* deliver before 160 minutes following the loading dose
* require rescue boluses in the first 80 minutes after initiation of PIEB (that is, before the 2nd PIEB bolus)
* withdraw their consent.

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: Women admitted to the Labor and Delivery unit at Mount Sinai Hospital that request to receive epidural analgesia.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Change in Lower sensory block level over time | 20 to 160 minutes post-loading dose
  The lower sensory block level to ice, defined as the dermatome at which there is a complete loss of cold perception. This will be measured at 20, 60, 80, 90, 100, 110, 120, 130, 140, 150, and 160 minutes post-loading dose of epidural medication.
Change in Upper sensory block level over time | 20 to 160 minutes post-loading dose
  The upper sensory block level to ice is defined as the dermatome at which there is an altered cold perception without complete sensitivity loss. This will be measured at 20, 60, 80, 90, 100, 110, 120, 130, 140, 150, and 160 minutes post-loading dose of epidural medication.

SECONDARY OUTCOMES:
Motor block score using Bromage score | 20 to 160 minutes post-loading dose
  Motor block will be assessed with the Bromage score: 0 = able to raise the extended leg; 1 = unable to raise the extended leg but able to flex knees; 2 = unable to flex knees, but able to flex ankle; 3 = unable to flex ankle. This will be measured at 20, 60, 80, 90, 100, 110, 120, 130, 140, 150, and 160 minutes post-loading dose of epidural medication.
Pain score | 20 to 160 minutes post-loading dose
  Pain score using verbal numerical rating scale (VNRS) (0-10, where 0=no pain and 10=worst pain ever). This will be measured at 20, 60, 80, 90, 100, 110, 120, 130, 140, 150, and 160 minutes post-loading dose of epidural medication.
Additional analgesia administered | 160 minutes
  Use and timing of use of PCEA and/or manual bolus will be recorded if they are administered at any time during the study time period.

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casellato JF, Ye XY, Downey K, Carvalho JCA. Changes in sensory block level during a programmed intermittent epidural bolus regimen for labour analgesia: a prospective observational cohort study. Can J Anaesth. 2022 Dec;69(12):1471-1476. doi: 10.1007/s12630-022-02318-w. Epub 2022 Sep 8. PMID 36076123